CLINICAL TRIAL: NCT04220801
Title: A Randomized, Double-blind, Placebo-controlled, Sequential Single and Multiple Ascending Dose (SAD/MAD) Study Following Oral Administration in Healthy Subjects to Evaluate the Safety, Tolerability, and Pharmacokinetics of ZM-H1505R
Brief Title: A Study of Orally Administered ZM-H1505R to Evaluate Safety, Tolerability and Pharmacokinetics After Single and Multiple Ascending Doses in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Zhimeng Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: ZM-H1505R-101
Record Dates: First submitted 2019-12-23; First posted 2020-01-07 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1 of Part 1 (SAD) (Experimental): 300 mg ZM-H1505R or placebo
  Interventions: Drug: ZM-H1505R
- Cohort 2 of Part 1(SAD) (Experimental): 450 mg ZM-H1505R or placebo
  Interventions: Drug: ZM-H1505R
- Cohort 3 of Part 1(SAD) (Experimental): 150 mg ZM-H1505R or placebo (2 periods)
  Interventions: Drug: ZM-H1505R
- Cohort 4 of Part 1(SAD) (Experimental): 75 mg ZM-H1505R or placebo
  Interventions: Drug: ZM-H1505R
- Cohort 5 of Part 1(SAD) (Experimental): 25 mg ZM-H1505R or placebo
  Interventions: Drug: ZM-H1505R
- Cohort 1 of Part 2 (MAD) (Experimental): 75 mg ZM-H1505R or placebo
  Interventions: Drug: ZM-H1505R
- Cohort 2 of Part 2 (MAD) (Experimental): 150 mg ZM-H1505R or placebo
  Interventions: Drug: ZM-H1505R
- Cohort 3 of Part 2 (MAD) (Experimental): 300 mg ZM-H1505R or placebo
  Interventions: Drug: ZM-H1505R

INTERVENTIONS:
Drug: ZM-H1505R — Single oral doses of 300, 450, 600, 750, and 900 mg of ZM-H1505R or placebo and multiple oral doses of 450, 600, and 750 mg of ZM-H1505R or placebo will be administered in a fasted state, or in the case of Cohort 3 (Part 1), a second dose of 600 mg will be administered in the fed state. During each SAD and MAD dosing period, 2 subjects in each cohort will receive placebo instead of ZM-H1505R. The dose levels may be adjusted based on the safety and tolerability obtained from the previous cohort.

SUMMARY:
ZM-H1505R is an investigational drug developed by Shanghai Zhimeng Biopharma Inc. for the treatment of Chronic Hepatitis B.

The purpose of this study is to see how safe the study drug is and how well it is tolerated after dosing. The study will also test how the study drug is taken up and eliminated by the body. An additional part of the study is to look at how this could be changed by giving the study drug with food.

ELIGIBILITY:
Inclusion Criteria:

* 1. Are capable of giving informed consent and complying with study procedures;
* 2. Are between the ages of 18 and 55 years, inclusive;
* 3. Female subjects have a negative pregnancy test results at screening and Day -1, and meet one of the following criteria:

  1. Using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives) [e.g., hormonal contraceptives (oral, patch, injectable or vaginal ring), implantable device (implantable rod or intrauterine device), or a double barrier (e.g., diaphragm, cervical cap, oral, patch or vaginal hormonal contraceptive, condom, spermicide, or sponge)]
  2. Surgically sterile for at least 3 months prior to screening by one of the following means:

     * Bilateral tubal ligation
     * Bilateral salpingectomy (with or without oophorectomy)
     * Surgical hysterectomy
     * Bilateral oophorectomy (with or without hysterectomy)
  3. Postmenopausal, defined as the following:

     * Last menstrual period greater than 12 months prior to screening
     * Postmenopausal status confirmed by serum FSH and estradiol levels at screening;
* 4. Considered healthy by the Investigator, based on subject's reported medical history, full PE, clinical laboratory tests, 12-lead ECG, and vital signs;
* 5. Normal liver function (AST/ALT < 1.5x ULN) and normal renal function (eGFR> 60mL/min/1.73 m2) as determined by Investigator following review of clinical laboratory test results;
* 6. Non-smoker and no nicotine containing products (including e-cigarettes) within 6 months;

  -- 7. Body mass index (BMI) of 18.0 to 32.0 kg/m2 inclusive and body weight not less than 50 kg;
* 8. Willing and able to adhere to study restrictions and to be confined at the clinical research center.
* 9. Male subjects with female partners of child bearing potential must agree to use condoms for the duration of the study and until 12 weeks after dosing with the study drug and must refrain from donating sperm for this same period.

Exclusion Criteria:

* 1. Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity as determined by the Investigator;
* 2. Reported or suspected malignancy;
* 3. Reported history of pancreatitis or gall stones;
* 4. Reported history of unexplained syncope, symptomatic hypotension or hypoglycemia;
* 5. Reported family history of long QTc syndrome;
* 6. Reported history of chronic diarrhea, malabsorption, unexplained weight loss, food allergies or intolerance;
* 7. Poor venous access;
* 8. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibody;
* 9. Donated or lost >500ml of blood in the previous 3 months;
* 10. Taken an investigational drug or participated in a clinical trial within 3 months (or 5 half-lives), whichever is longer;
* 11. Taken any prescription medications within 14 days or 5 half-lives (whichever is longer) of the first dose of study drug;
* 12. Hospital admission or major surgery within 6 months prior to screening;
* 13. A reported history of prescription drug abuse, or illicit drug use within 9 months prior to screening;
* 14. A reported history of alcohol abuse according to medical history within 9 months prior to screening;
* 15. A positive screen for alcohol, drugs of abuse at screening or Day -1;
* 16. An unwillingness or inability to comply with food and beverage restrictions during study participation;
* 17. Use of over-the-counter (OTC) medication within 7 days, and herbal supplements (including St John's Wort, herbal teas, garlic extracts) within 7 days prior to dosing (Note: Use of acetaminophen at < 2 g/day is permitted until 24 hours prior to dosing)
* 18. Any condition or finding that in the Investigators opinion would put the subject or study conduct at risk if the subject were to participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events and Serious Adverse Events | 22 days for Cohorts 1, 2, 4, and 5; 36 days for Cohort 3 in part 1 and Chorts in part 2
  Safety data from subjects in Part 1 and Part 2 treated with placebo will be pooled, respectively.
  Safety evaluations will be based on the incidence, intensity, and relatedness of AEs
Number of Participants With Abnormal Physical Examinations | 22 days for Cohorts 1, 2, 4, and 5; 36 days for Cohort 3 in part 1 and Chorts in part 2
  Safety data from subjects in Part 1 and Part 2 treated with placebo will be pooled, respectively.
  Safety evaluations will be based on the incidence, intensity, and relatedness of AEs and changes in subject PE findings
Number of Participants With Abnormal Vital Signs | 22 days for Cohorts 1, 2, 4, and 5; 36 days for Cohort 3 in part 1 and Chorts in part 2
  Safety data from subjects in Part 1 and Part 2 treated with placebo will be pooled, respectively.
  Safety evaluations will be based on the incidence, intensity, and relatedness of AEs and changes in subject vital signs
Number of Participants With Clinically Significant Laboratory Findings | 22 days for Cohorts 1, 2, 4, and 5; 36 days for Cohort 3 in part 1 and Chorts in part 2
  Safety data from subjects in Part 1 and Part 2 treated with placebo will be pooled, respectively.
  Safety evaluations will be based on the incidence, intensity, and relatedness of AEs and changes in subject clinical laboratory results
Number of Participants With Abnormal ECGs | 22 days for Cohorts 1, 2, 4, and 5; 36 days for Cohort 3 in part 1 and Chorts in part 2
  Safety data from subjects in Part 1 and Part 2 treated with placebo will be pooled, respectively.
  Safety evaluations will be based on the incidence, intensity, and relatedness of AEs and changes in subject ECGs.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Tracey, MD., Principal Investigator — Frontage Clinical Services, Inc.
Locations (1):
- Frontage Clinical Services, Secaucus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang X, Hua B, Liu G, Xia T, Deng A, Lu H, Guo R, Wang Z, Liang B, Chen H, Jin Q, Zhang Z. Safety, Tolerability, and Pharmacokinetics of a Novel Human Hepatitis B Virus Capsid Assembly Modulator Canocapavir: A Randomized First-in-Human Study. Gastro Hep Adv. 2023 Jan 7;2(4):524-531. doi: 10.1016/j.gastha.2023.01.001. eCollection 2023. PMID 39132049